CLINICAL TRIAL: NCT07104513
Title: Study on the Long-term Efficacy Evaluation and Influencing Factors of Repeated Low-level Red-light Therapy in Myopia Prevention and Control in Children
Brief Title: Efficacy and Influencing Factors of Repeated Low-level Red-light in Myopia
Acronym: RLRL
Status: Active, not recruiting | Type: Observational
Sponsor: Ruihua Wei (Other)
Responsible Party: Sponsor-Investigator, Ruihua Wei, Professor, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Other Study IDs: 2025KY-41
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- The RLRL-1year Group: use red light 1 year
  Interventions: Device: Red Light
- The RLRL-2years Group
  Interventions: Device: Red Light
- The RLRL-3years Group
  Interventions: Device: Red Light
- The RLRL-more than 3 years: use the RLRL-more than 3 years
  Interventions: Device: Red Light

INTERVENTIONS:
Device: Red Light — use red light twice per day, both eyes. use red light for one year in The RLRL-1year Group. use red light for two year in The RLRL-2years Group. red light for three years in The RLRL-3years Group.red light for more than three years in The RLRL- more than 3years Group.

SUMMARY:
To evaluate the long-term efficacy of repeated low-level red-light (RLRL) therapy in the prevention and control of myopia in children, and to analyze the key factors influencing its efficacy (such as individual differences and compliance), with the aim of providing evidence-based support for the optimization of clinical myopia prevention and control strategies.

DETAILED DESCRIPTION:
This is a real world multi-centre study. The devices are connected to the internet with an automated diary function to record treatment sessions and to monitor patient compliance.The total sample size of 3000 arerandomly allocated into treatment groups,observation for 1 year and more.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 5 to 16, gender unrestricted;
2. RLRL device usage duration of one year or more.

Exclusion Criteria:

* Children with obvious strabismus and amblyopia
* With congenital eye disease, such as congenital cataract, congenital retinal disease
* Secondary myopia (such as premature retinopathy or other eye diseases in infants and children caused secondary myopia), or myopia combined with systemic syndrome (such as Marfan syndrome)
* Had internal eye surgery (such as cataract extraction, intraocular lens implantation, anti-glaucoma surgery, etc.)
* Refractive medium opacity (such as corneal disease, crystal opacity, etc.)
* Bnormal intraocular pressure and clinical significance (IOP <10 mmHg or IOP >21mmHg or binocular IOP difference ≥5mmHg)
* Fundus chorioretinopathy (except for high myopia fundus degenerative changes) or other intraocular diseases
* Optic nerve damage or congenital optic nerve dysfunction
* Can not be regularly checked
* The adjustment range is less than 8D or obvious near difficulties
* Other reasons researchers think it is not suitable for inclusion in researchers

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 5-16 years old, 500
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-09-28 (Actual); Primary Completion 2028-07-28 (Estimated); Study Completion 2030-07-28 (Estimated)

PRIMARY OUTCOMES:
axial length | up to 72 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Eye Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No